CLINICAL TRIAL: NCT02953873
Title: Dosing Requirements of Astagraf XL® in African American Kidney Transplant Recipients Converted From Twice-daily Tacrolimus
Brief Title: Dosing Requirements of Astagraf XL® in African American Kidney Transplant Recipients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: Astellas Pharma Inc (Industry)
Responsible Party: Principal Investigator, James N. Fleming, Principal Investigator, Medical University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00061221
Record Dates: First submitted 2016-11-01; First posted 2016-11-03 (Estimated); Results first posted 2019-12-26 (Actual); Last update posted 2019-12-26 (Actual); Status verified 2019-12

CONDITIONS: Immunosuppression
MeSH Terms: interventions — Tacrolimus; Mycophenolic Acid; Prednisone; Adrenal Cortex Hormones; Methylprednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Conversion Arm (Other): Tacrolimus Extended Release Capsule (goal 5 - 12ng/mL) + Mycophenolate Mofetil ≥500mg twice a day OR Mycophenolate Sodium ≥360mg twice a day+ prednisone ≥ 5mg Daily
  Interventions: Drug: Tacrolimus Extended Release Capsule; Drug: Mycophenolate mofetil; Drug: Prednisone; Drug: Mycophenolate Sodium

INTERVENTIONS:
Drug: Tacrolimus Extended Release Capsule — goal trough 5 - 12ng/mL
  Other Names: Astagraf XL
Drug: Mycophenolate mofetil — ≥500mg twice a day
  Other Names: Cellcept
Drug: Prednisone — goal dose 5mg daily
  Other Names: Corticosteroids; Methylprednisolone
Drug: Mycophenolate Sodium — ≥360mg twice a day
  Other Names: Myfortic

SUMMARY:
Compare the difference in dose-normalized trough and total daily dose necessary to reach the steady state therapeutic goal after conversion from tacrolimus IR to Astagraf XL® in African American kidney transplant recipients.

DETAILED DESCRIPTION:
The purpose of this study is to compare the difference in medication dosage and total daily dose necessary of Astagraf XL® in order to reach therapy goal, when taken with other medications that are routinely used for kidney transplantation, which may stop the development of a substance that can cause long-term damage to the transplanted kidney. African American kidney transplant patients aged 18 and above who are underwent a kidney transplant are eligible to participate. The duration of the study is 3 months.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age
2. Signed informed consent
3. African American race
4. History of a solitary renal transplant
5. Stable tacrolimus dose for at least 2 weeks prior to randomization

Exclusion Criteria:

1. A condition or disorder that, in the opinion of the investigator, may adversely affect the outcome of the study or the safety of the subject
2. Currently enrolled in an investigational drug trial
3. History of a non-renal organ transplant
4. History of acute cellular rejection within 1 month prior to randomization
5. An increase in serum creatinine by > 20% in the 2 weeks prior to randomization
6. Maintenance immunosuppression that does not consist of tacrolimus IR given twice daily, mycophenolate mofetil > 1000mg TDD or mycophenolate sodium > 720mg TDD, and prednisone ≥ 5mg daily

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-05-05 (Actual); Primary Completion 2018-09-10 (Actual); Study Completion 2018-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Fleming, PharmD, Principal Investigator — Medicual U of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No
The data will not be shared.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Conversion Arm
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Conversion Arm
Number analyzed (Participants) | 25
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 52 [40 to 58]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 25
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Number of Days Since Transplant [Median (Inter-Quartile Range); unit: days] | 270 [202 to 496]
Weight [Mean (Standard Deviation); unit: kilograms] | 94.5 (23)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 31.7 (6.1)
Calculated Panel Reactive Antibodies (cPRA) [Median (Inter-Quartile Range); unit: percent] — Calculated Panel Reactive Antibodies (cPRA) is used to determine the likelihood that a transplant recipient and donor would be incompatible. The scale goes from 0% to 100 %. A higher % means there is a higher likelihood that the recipient and donor are incompatible.
  percent | 50 [5 to 79]
Number of participants on Hemodialysis Prior to Transplant [Count of Participants; unit: Participants] | 23
Cold Ischemic Time [Median (Inter-Quartile Range); unit: hours] — The Cold Ischemic Time is the amount of time that the donor kidney has blood supply cut off. The time starts when blood supply is cut off from the donor kidney and put on ice, and ends when the kidney is taken out of ice in preparation for transplant to the recipient.
  hours | 18.1 [10.1 to 25.1]
Warm Ischemic Time [Mean (Standard Deviation); unit: minutes] — The warm ischemia time is the amount of time, from when the donor kidney is taken out of ice until the kidney has blood flow restored in the transplant recipient.
  minutes | 38.7 (7.1)

OUTCOME MEASURES:

1. Primary Outcome: Dose-normalized Trough
Description: Difference in dose-normalized trough at steady state before and after conversion from tacrolimus IR to Astagraf XL®
Time Frame: Baseline to 3 months post-conversion
Measure: Median (Inter-Quartile Range); unit: ng/dL
Arm/Group | Conversion Arm
Number analyzed (Participants) | 25
ng/dL
  Pre-Conversion Dose Trough | 0.59 [0.50 to .76]
  Post-Conversion Dose Trough | 0.44 [0.39 to 0.80]

2. Secondary Outcome: Total Daily Dose
Description: Difference in Total Daily Dose necessary for steady state therapeutic goal
Time Frame: Baseline to 3 months post conversion
Measure: Median (Inter-Quartile Range); unit: mg
Arm/Group | Conversion Arm
Number analyzed (Participants) | 25
mg
  Pre-Conversion Tacrolimus Dose | 10 [9 to 17]
  Post-Conversion Tacrolimus Dose | 15 [10 to 17.5]

3. Secondary Outcome: Weight-Based Dose Requirement
Description: Weight-based dose requirements to reach therapeutic goal pre- and post-conversion
Time Frame: Baseline to 3 months post conversion
Measure: Median (Inter-Quartile Range); unit: mg/kg
Arm/Group | Conversion Arm
Number analyzed (Participants) | 25
mg/kg
  Pre-Conversion | 0.11 [0.10 to 0.17]
  Post-Conversion | 0.16 [0.11 to 0.20]

4. Secondary Outcome: Number of Days to Reach Therapeutic Trough Goal
Description: Days to reach therapeutic goal after conversion
Time Frame: Baseline to 3 months post conversion
Population: Days to reach therapeutic goal was further separated by CYP3A5 1 expression.
Measure: Median (Inter-Quartile Range); unit: number of days
Arm/Group | Conversion Arm
Number analyzed (Participants) | 25
number of days
  Homozygous CYP3A5 1 expressors: number analyzed (Participants) | 12
  Homozygous CYP3A5 1 expressors | 15 [5 to 25]
  Heterozygous CYP3A5 1 expressors: number analyzed (Participants) | 10
  Heterozygous CYP3A5 1 expressors | 10 [5 to 15]
  CYP3A5 1 non-expressors: number analyzed (Participants) | 3
  CYP3A5 1 non-expressors | 15 [15 to 15]

5. Secondary Outcome: Dose Modifications
Description: Number of dose modifications from baseline to 3 months post-conversion.
Time Frame: Baseline to 3 months post conversion
Population: 12 participants are homozygous, 10 are heterozygous, and 3 are non-expressors. This represents the 25 total subjects in the study.
Measure: Median (Inter-Quartile Range); unit: number of dose modifications
Arm/Group | Conversion Arm
Number analyzed (Participants) | 25
number of dose modifications
  Homozygous CYP3A5 1 expressors: number analyzed (Participants) | 12
  Homozygous CYP3A5 1 expressors | 1 [0 to 3]
  Heterozygous CYP3A5 1 expressors: number analyzed (Participants) | 10
  Heterozygous CYP3A5 1 expressors | 2 [0 to 2]
  CYP3A5 1 non expressers: number analyzed (Participants) | 3
  CYP3A5 1 non expressers | 4 [1 to NA] — The value is not applicable. There were only 3 values in the non-expressers, so a 75% interquartile range is not applicable.

ADVERSE EVENTS:
Time Frame: Adverse events were collected over 3 months
Arm/Group | Conversion Arm
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 1/25
Other Adverse Events (participants affected / at risk) | 19/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Conversion Arm (N=25)
Chronic myeloid Leukemia (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Conversion Arm (N=25)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3)
Pain (General disorders) | 5 (5)
Bleeding (Blood and lymphatic system disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Skin infection (abscess) (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperglycemia (Endocrine disorders) | 2 (2)
Gait disturbance (General disorders) | 1 (1)
Headache (General disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Urinary Tract Infection (Renal and urinary disorders) | 1 (1)
Muscle Myositis (Musculoskeletal and connective tissue disorders) | 1 (1)
Chronic myeloid leukemia (Blood and lymphatic system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-12): https://cdn.clinicaltrials.gov/large-docs/73/NCT02953873/Prot_SAP_000.pdf